CLINICAL TRIAL: NCT02268084
Title: A Randomized Double-Blind Placebo-Controlled Trial to Evaluate Treatment Efficacy of EEG/ECD-Guided Magnetic Resonant Therapy in Combat Veterans With Post-Traumatic Stress Disorder (PTSD).
Brief Title: Trial to Evaluate Efficacy of Magnetic Resonant Therapy (MRT) in PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wave Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRT-002
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Results first posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; TMS; EEG
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Sham controlled
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Stimulation (Sham Comparator): Sham treatment will consist of 6 seconds a minute for 30 minutes a day, 5 days a week for 2 weeks (double blind phase only) using a sham device. Sham device mimics the same noise and sensation of active treatment.
  Interventions: Device: Sham
- Active sTMS (Active Comparator): Active treatment will consist of 6 seconds a minute for 30 minutes a day, 5 days a week for 2 weeks (double blind phase) and 2 additional weeks for all subjects (open label) with Synchronized Transcranial Magnetic Stimulation (sTMS), using an active device.
  Interventions: Device: Magnetic EEG/ECG-guided Resonance Therapy

INTERVENTIONS:
Device: Magnetic EEG/ECG-guided Resonance Therapy — A coil delivers a pulsed magnetic field to the cortex of the brain
  Other Names: Magnetic Resonant Therapy; Magnetic e-Resonance Therapy; MeRT; MRT
  Arms: Active sTMS
Device: Sham — Sham coil simulates behavior of the intervention magnetic coil without applying the magnetic field
  Arms: Sham Stimulation

SUMMARY:
The purpose of this study is to establish the efficacy of Magnetic Resonant Therapy in treating Post Traumatic Stress Disorder in Veterans.

DETAILED DESCRIPTION:
This clinical trial is a prospective, randomized, double-blinded, placebo-controlled study designed to evaluate the safety and efficacy of EEG/ECG-guided magnetic resonant therapy (MRT) in combat veterans with Posttraumatic Stress Disorder. A total of 2004 subjects will be treated in two phases: double-blind and open label.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to adhere to the treatment schedule and all required study visits.
* Any non-Active Duty Military are included.
* PCL-M > 45
* Primary diagnosis of Posttraumatic Stress Disorder rendered by the Clinician Administered PTSD Scale (CAPS)

Exclusion Criteria:

* Individuals diagnosed by the Investigator with the following conditions (current unless otherwise stated): History of open skull traumatic brain injury. History of clinically significant seizure disorder.
* Individuals with a clinically defined neurological disorder including, but not limited to: Any condition likely to be associated with increased intracranial pressure. Space occupying brain lesion. History of cerebrovascular accident. Cerebral aneurysm.
* EEG abnormalities that indicate risk of seizure, i.e., abnormal focal or general slowing or spikes during the EEG recording.
* Any type of rTMS treatment within 3 months prior to the screening visit.
* Currently under antipsychotic medication treatment.
* Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, stents, or electrodes) or any other metal object within or near the head, excluding the mouth, which cannot be safely removed.
* Clinically significant abnormality or clinically significant unstable medical condition that in the Investigator's judgment might pose a potential safety risk to the subject or limit interpretation of the trial results.
* Clinically significant medical illness, including any uncontrolled thyroid disorders, hepatic, cardiac, pulmonary and renal malfunctioning.
* Any condition which in the judgment of the investigator would prevent the subject from completion of the study.
* Inability to acquire a clinically satisfactory EEG/ECG on a routine basis.
* Grossly abnormal electrolyte or cell blood count panels suggestive of other pathology at study initiation.
* Active Duty Military are excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Tahgva, MD, Principal Investigator — 8583607260
Locations (1):
- Del Mar Center for Neurorestoration, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were screened for eligibility; subjects with history of seizure disorder, history of intracranial lesion, history of intracranial implant, prior transcranial magnetic therapy, and inability to adhere to the treatment schedule were excluded from the study. Eligible subjects were provided with study consent forms. No medication wash-out was required.
Groups:
- Active: Magnetic EEG/ECG-Guided Resonance Therapy treatments use a coil to deliver pulsed magnetic fields to the cortex of the brain. Active treatments are administered for 6 seconds/minute for 30 minutes/day, 5 days/week for four weeks (two weeks of double-blind treatment, two weeks of open-label treatment).
- Sham: Sham treatment devices simulate the behavior of the active devices by mimicking the same noise and sensation of active treatment without applying the magnetic field. Sham treatments are administered for 6 seconds/minute for 30 minutes/day, 5 days/week for two weeks. Active treatment devices were used for the additional 2 weeks of open-label treatment.
Period: Overall Study
Arm/Group | Active | Sham
Started | 49 | 47
Completed | 40 | 40
Not Completed | 9 | 7
Not completed — Three subjects in the sham had early blind code opening due to symptomatic worsening. | 0 | 3
Not completed — Combination of the following, exact numbers not available: Lost to follow-up, voluntary withdrawal | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Sham: Shame treatment devices simulate the behavior of the active devices by mimicking the same noise and sensation of active treatment without applying the magnetic field. Sham treatments are administered for 6 seconds/minute for 30 minutes/day, 5 days/week for two weeks. Active devices were used for the additional two weeks of open-label treatment.
- Total: Total of all reporting groups
Arm/Group | Active | Sham | Total
Number analyzed (Participants) | 49 | 47 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 47 | 96
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender data unavailable for overall population.
  Participants
    number analyzed (Participants) | 40 | 40 | 80
    Female | 3 | 5 | 8
    Male | 37 | 35 | 72
Region of Enrollment [Number; unit: participants]
  United States | 49 | 47 | 96

OUTCOME MEASURES:

1. Primary Outcome: Mean (SD) Change in Post-Traumatic Stress Disorder Checklist - Military Version (PCL-M) Scores From Baseline to End of Double-Blind Phase
Description: Mean change in the PCL-M total scores of subjects from baseline to end of the double-blind treatment phase, compared between active and sham groups.
  The Post-traumatic Stress Disorder Checklist - Military Version (PCL-M) is a 17-item metric for PTSD symptoms, as defined by the DSM-IV. Each symptom is scored on a scale from 1-5; total scores range from 17 (least symptomatic) to 85 (most symptomatic).
Time Frame: Baseline (Day 0) and End of Double-Blind Treatment (Week 2)
Population: 96 participants were randomized into the trial, 86 completed treatment protocol. Of those, 6 were excluded from final analyses for failing to meet protocol requirements. Analyses were performed on the remaining 80 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active: Magnetic EEG-Guided Resonance Therapy Treatments use a coil to deliver pulsed magnetic fields to the cortex of the brain. Active treatments are administered for 6 seconds/minute for 30 minutes/day, 5 days/week for four weeks (two weeks of double blind treatment, two weeks of open-label treatment.
- Sham: Sham treatment devices simulate the behavior of the active devices by mimicking the same noise and sensation of active treatment without applying the magnetic field. Sham treatments are administered for 6 seconds/minute for 30 minutes/day, 5 days/week for two weeks. Active devices were used for the additional two weeks of open-label treatment.
Arm/Group | Active | Sham
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 65.78 (9.71) | 65.25 (8.87)
  Change Between Baseline and Week 2 | -22.45 (14.70) | -14.75 (16.56)
Statistical Analysis 1: Comparison: Active vs Sham; Null hypothesis is that the active treatment group does not differ from the sham group in changes in the PCL-M total scores; Test type: Superiority; p = .007, ANOVA

2. Secondary Outcome: Mean (SD) Change in Post-Traumatic Stress Disorder Checklist - Military Version (PCL-M) Scores From Baseline to End of Open-Label Treatment Phase
Description: Mean change in the PCL-M total scores of subjects from baseline to end of the open-label treatment phase, compared between active and sham groups.
  The Post-traumatic Stress Disorder Checklist - Military Version (PCL-M) is a 17-item metric for PTSD symptoms, as defined by the DSM-IV. Each symptom is scored on a scale from 1-5; total scores range from 17 (least symptomatic) to 85 (most symptomatic).
Time Frame: Baseline (Day 0) and End of Open-Label Treatment (Week 4)
Population: 96 participants were randomized into the trial, 86 completed treatment protocol. Of those, 6 were excluded from final analyses for failing to meet the protocol requirements. Analyses were performed on the remaining 80 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active: Magnetic EEG-Guided Resonance Therapy treatments use a coil to deliver pulsed magnetic fields to the cortex of the brain. Active treatments are administered for 6 seconds/minute for 30 minutes/day, 5 days/week for four weeks.
  Active group received two weeks of active treatment in the double-blind phase, and two weeks in the open-label treatment.
- Sham: Sham treatment devices simulate the behavior of the active devices by mimicking the noise and sensation of active treatment without applying the magnetic field. Sham treatments are administered for 6 seconds/minute for 30 minutes/day, 5 days/week for two weeks.
  Sham group received two weeks of sham treatment in the double-blind phase, and two weeks of active treatment in the double-blind phase.
Arm/Group | Active | Sham
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 65.78 (9.71) | 65.25 (8.87)
  Change from Baseline to Week 4 (End of Open-Label) | -32.53 (13.07) | -30.9 (13.34)
Statistical Analysis 1: Comparison: Active vs Sham; Test type: Superiority; p = .326, t-test, 2 sided

3. Secondary Outcome: Mean (SD) Change in Pittsburgh Sleep Quality Index - Addendum for PTSD (PSQI-A) Score From Baseline to End of Double-Blind Treatment
Description: Mean change in the PSQI-A total scores from baseline to end of the double-blind treatment, compared between active and sham groups.
  The Pittsburgh Sleep Quality Index - Addendum for PTSD (PSQI-A) is a 7-item metric to rate sleep disturbance items that are commonly reported with PTSD. Total scores range from 0 (least severe) to 21 (most severe), where scores greater than or equal to 4 have been used to identify adults with PTSD.
Time Frame: Baseline (Day 0) and End of Double-Blind Treatment (Week 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active: Magnetic EEG-Guided Resonance Therapy treatments use a coil to deliver pulsed magnetic fields to the cortex of the brain. Active treatments are administered for 6 seconds/minute for 30 minutes/day, 5 days/week for four weeks (two weeks of double-blind treatment, two weeks of open-label treatment).
- Sham: Sham treatment devices simulate the behavior of the active devices by mimicking the same noise and sensation of active treatment without applying the magnetic field. Sham treatments are administered for 6 seconds/minute fro 30 minutes/day, 5 days/week for two weeks. Active devices were used for the additional two weeks of open-label treatment.
Arm/Group | Active | Sham
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 10.85 (4.95) | 9.67 (4.67)
  Change Between Baseline and Week 2 | -4.66 (5.54) | -2.03 (4.48)

4. Secondary Outcome: Mean (SD) Change in Pittsburgh Sleep Quality Index - Addendum for PTSD (PSQI-A) Score From Baseline to End of Open-Label Treatment
Description: Mean change is the PSQI-A total scores from baseline to end of the open-label treatment, compared between active and sham groups.
  The Pittsburgh Sleep Quality Index - Addendum for PTSD (PSQI-A) is a 7-item metric to rate sleep disturbance items that are commonly reported with PTSD. Total scores ranges from 0 (least severe) to 21 (most severe), where scores greater than or equal to 4 have been used to identify adults with PTSD.
Time Frame: Baseline (Day 0) and End of Open-Label Treatment (Week 4)
Population: 96 participants were randomized into the trial, 86 completed treatment protocol. Of those, 6 were excluded from the final analyses for failing to meet the protocol requirements. Analyses were performed on the remaining 80 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Sham
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 10.84 (4.95) | 9.67 (4.67)
  Change from Baseline to Week 4 (End of Open-Label) | -7.23 (5.40) | -5.39 (4.74)

5. Secondary Outcome: Mean (SD) Change in Hamilton Depression Rating Scale (HAMD-17) Scores From Baseline to End of Double-Blind Treatment
Description: Mean change in the HAMD-17 total scores from baseline to end of double-blind treatment, compared between active and sham
  The Hamilton Depression Rating Scale (HAMD-17) is a 17-item metric to rate subjects on severity of depressive symptoms. Total scores range from 0-52, with higher scores indicating more severe symptoms; a score of 0-7 is generally accepted to be within normal range (or in remission), while a score of 20 or greater indicates moderate to severe depression.
Time Frame: Baseline (Day 0) and End of Double-Blind Treatment (Week 2)
Population: 96 participants were randomized into the trial, 86 completed treatment protocol. Of those, 6 were excluded from the final analyses for failling to meet the protocol requirements. Analyses were performed on the remaining 80 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active: Magnetic EEG-Guided Resonance Therapy treatments use a coil to deliver pulsed magnetic fields to the cortex of the brain. Active treatments are administered for 6 seconds/minute for 30 minutes/day, 5 days/week for four weeks (two weeks of double-blind treatment, two weeks of open label treatment).
- Sham: Sham treatment devices simulate the behavior of the active devices by mimicking the same noise and sensation of the active treatment without applying the magnetic field. Sham treatments are administered for 6 seconds/minute for 30 minutes/day, 5 days/week for two weeks. Active devices were used for the additional two weeks of open-label treatment.
Arm/Group | Active | Sham
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 24.23 (8.01) | 22.55 (8.25)
  Change Between Baseline and Week 2 | -11.33 (1.77) | -8.08 (.02)

6. Secondary Outcome: Mean (SD) Change in Hamilton Depression Rating Scale (HAMD-17) Scores From Baseline to End of Open-Label Treatment
Description: Mean change in the HAMD-17 total scores from baseline to end of open-label treatment, compared between active and sham groups.
  The Hamilton Depression Rating Scale (HAMD-17) is a 17-item metric to rate subjects on severity of depressive symptoms. Total scores range from 0-52, with higher scores indicating more severe symptoms; a score of 0-7 is generally accepted to be within normal range (or in remission), while a score of 20 or greater indicates moderate to severe depression.
Time Frame: Baseline (Day 0) and End of Open-Label Treatment (Week 4)
Population: 96 participants were randomized into the trial, 86 completed treatment protocol. Of those, 6 were excluded from the final analyses for failing to meet protocol requirements. Analyses were performed on the remaining 80 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Sham
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 24.23 (8.01) | 22.55 (8.25)
  Change from Baseline to Week 4 (End of Open-Label) | -16.60 (2.40) | -15.43 (2.00)

7. Secondary Outcome: Mean (SD) Change in World Health Organization's Quality of Life Index (WHO-QOL) Domain Scores From Baseline to End of Treatment
Description: Mean change in each WHO-QOL domain score from baseline to end of treatment, compared between active and sham groups.
  The World Health Organization's Quality of Life Index - BREF Version (WHO-QOL) is a metric used to establish the subject's quality of life in four domains: physical health (D1), psychological health (D2), social relationships (D3), and environmental health (D4). Higher scores indicate a more positive quality of life; D1 has a score range of 7-35, D2 has a range of 6-30, D3 has a range of 3-15, D4 has a range of 8-40.
Time Frame: Baseline and End of Double-Blind (Week 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Sham
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline (D1) | 18.89 (2.87) | 18.28 (2.67)
  Change Between Baseline and Week 2 (D1) | 3.11 (3.82) | 1.59 (4.90)
  Baseline (D2) | 16.18 (2.71) | 17.03 (3.60)
  Change Between Baseline and Week 2 (D2) | 2.63 (3.74) | 0.97 (2.96)
  Baseline (D3) | 7.36 (2.78) | 7.82 (2.46)
  Change Between Baseline and Week 2 (D3) | 1.89 (2.73) | 1.59 (2.10)
  Baseline (D4) | 27.00 (5.01) | 30.74 (5.86)
  Change Between Baseline and Week 2 (D4) | 2.76 (3.89) | 0.56 (3.31)

8. Secondary Outcome: Mean (SD) Change in World Health Organization's Quality of Life Index (WHO-QOL) Domain Score From Baseline to End of Open-Label Treatment
Description: Mean change in each WHO-QOL domain score from baseline to end of open-label treatment, compared between active and sham groups.
  The World Health Organization's Quality of Life Index - BREF Version (WHO-QOL) is a metric used to establish the subject's quality of life in four domains: physical health (D1), psychological health (D2), social relationships (D3), and environmental health (D4). Higher scores indicate a more positive quality of life; D1 has a score range of 7-35, D2 has a range of 6-30, D3 has a range of 3-15, D4 has a range of 8-40.
Time Frame: Baseline (Day 0) and End of Open-Label (Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Sham
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline (D1) | 18.89 (2.82) | 18.28 (2.67)
  Change from Baseline to Week 4 (End of Open-Label) (D1) | 5.56 (3.54) | 4.83 (3.30)
  Baseline (D2) | 16.18 (2.71) | 17.02 (3.60)
  Change from Baseline to Week 4 (End of Open-Label) (D2) | 4.50 (4.21) | 3.20 (3.23)
  Baseline (D3) | 7.37 (2.78) | 7.82 (2.46)
  Change from Baseline to Week 4 (End of Open-Label) (D3) | 3.19 (2.67) | 2.86 (2.06)
  Baseline (D4) | 27.00 (5.01) | 30.74 (5.86)
  Change from Baseline to Week 4 (End of Open-Label) (D4) | 5.47 (3.71) | 2.83 (3.69)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from date of consent through 30 days of last treatment date, on each treatment or follow-up day.
Description: Adverse events were collected on every treatment and assessment visit through self-reporting and observation.
Groups:
- Sham: Sham treatment will consist of 6 seconds a minute for 30 minutes a day, 5 days a week for 2 weeks (double blind phase only). Sham treatment mimicks same noise and sensation of active treatment.
  Sham: Sham coil simulates behavior of the intervention magnetic coil without applying the magnetic field
- Active: Active treatment will consist of 6 seconds a minute for 30 minutes a day, 5 days a week for 2 weeks (double blind phase) and 2 additional weeks for all subjects (open label).
  Magnetic EEG/ECG-guided Resonance Therapy: A coil delivers a pulsed magnetic field to the cortex of the brain
Arm/Group | Sham | Active
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/49
Other Adverse Events (participants affected / at risk) | 1/47 | 4/49
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sham (N=47) | Active (N=49)
Headache (Mild) (General disorders) | 1 | 4

LIMITATIONS AND CAVEATS:
* Sham condition imperfect; the sham device inadvertently delivers some treatment through magnetically shielded coil and forehead stimulation
* Placebo effects may modulate brain regions and neural networks similar to active treatment; it is common for both sham and active groups to show clinical improvement
* Gender influences PTSD symptoms and severity and response to treatment/efficacy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No